CLINICAL TRIAL: NCT01379651
Title: Specific Oral Tolerance Induction in Children With Severe Egg Allergy: A Randomized Controlled Trial Using a 6 Months Protocol
Brief Title: Time-limited Specific Oral Tolerance Induction in Children With Severe Egg Allergy
Acronym: EGGSOTI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ospedale Buon Consiglio Fatebenefratelli (Other)
Responsible Party: Principal Investigator, Iride Dello Iacono, pediatrician, Ospedale Buon Consiglio Fatebenefratelli
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FBFBN
Record Dates: First submitted 2011-06-20; First posted 2011-06-23 (Estimated); Results first posted 2011-08-30 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: - Egg Hypersensitivity
Keywords: Egg allergy,specific oral tolerance induction
MeSH Terms: conditions — Egg Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Specific oral tolerance induction (Experimental): Specific oral tolerance induction consisted in the administration of increasing amounts of food antigen
  Interventions: Other: Specific oral tolerance induction
- control (No Intervention): controls were kept on an egg-free diet for 6 months

INTERVENTIONS:
Other: Specific oral tolerance induction — Specific oral tolerance induction consisted in the administration of increasing amounts of raw emulsion egg
  Other Names: SOTI
  Arms: Specific oral tolerance induction

SUMMARY:
To evaluate the efficacy of a 6-month specific oral tolerance induction (SOTI) protocol in inducing tolerance (maximal dose of raw egg emulsion tolerated) in children with severe IgE-mediated egg allergy and a history of at least 1 anaphylactic reaction after accidental exposure to egg.

DETAILED DESCRIPTION:
Oral immunotherapy consisted in the administration of increasing amounts of raw emulsion egg. The children started with 1 drop of undiluted raw egg emulsion (0.05 ml) flavored with vanilla and cacao, hidden by the parents in the child's breakfast (cow's milk, soymilk, fruit juice or other). The dose was doubled at intervals of about one month in the day hospital. The increases in dose were customized for each subject based on the frequency and severity of side effects, or when an inter-current illness or asthma worsening intervened during the SOTI.

The investigators limited the SOTI protocol to six months for all patients, irrespective of the dose reached, in order to favor the adherence of families to the study.

When objective symptoms seemed more important (grade 2, 3 and 4 reaction), medical treatment was given. Subjects were discontinued from the study in case of severe adverse reactions (grade 5 reaction). Parents were advised they could telephone investigators 24 hours a day

ELIGIBILITY:
Inclusion Criteria:

* at least 1 anaphylactic reaction (grade 3, 4 and 5 according to Sampson's grading after accidental exposure to trace amounts of egg or egg-derivative products, requiring emergency treatment, at least 1 year before enrollment
* demonstration of egg white specific IgE by the skin prick test (SPT), end-point SPT, raw egg white prick-by-prick (PP) and egg white-specific IgE determination
* positive double-blind placebo-controlled food challenge (DBPCFC) at a dose of less than 0.9 ml of raw emulsion egg

Exclusion Criteria:

* age below 5 years
* poorly controlled asthma
* parents with a history of unreliable management of complications and treatment.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iride Dello Iacono, pediatrician, Study Director — Unit of Pediatrics, Fatebenefratelli Hospital, Benevento, Italy
Locations (1):
- Unit of Pediatrics, Fatebenefratelli Hospital, Benevento, Benevento, Italy

REFERENCES:
- [Background] Calvani M, Giorgio V, Miceli Sopo S. Specific oral tolerance induction for food. A systematic review. Eur Ann Allergy Clin Immunol. 2010 Feb;42(1):11-9. PMID 20355360
- [Background] Sampson HA. Anaphylaxis and emergency treatment. Pediatrics. 2003 Jun;111(6 Pt 3):1601-8. PMID 12777599
- [Background] Sicherer SH, Sampson HA. 9. Food allergy. J Allergy Clin Immunol. 2006 Feb;117(2 Suppl Mini-Primer):S470-5. doi: 10.1016/j.jaci.2005.05.048. PMID 16455349
- [Background] Barbi E, Berti I, Longo G. Food allergy: from the of loss of tolerance induced by exclusion diets to specific oral tolerance induction. Recent Pat Inflamm Allergy Drug Discov. 2008 Nov;2(3):212-4. doi: 10.2174/187221308786241875. PMID 19076011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 26 children (14 boys, 12 girls; median age: 7 years 7 months; range 5-11 years), with severe IgE-mediated egg allergy (EA) were recruited from the Pediatric and Allergology Unit of the Fatebenefratelli Hospital in Benevento, Italy, from January 2008 to December 2009.
Pre-assignment Details: 6 children(4 males and 2 females)were excluded from the study: one child because the parents had a history of unreliable management of complications and treatments;2 children because of poorly controlled asthma;3 children because of a positive double-blind placebo-controlled food challenge (DBPCFC) at a dose of raw egg emulsion higher than 0.9 ml.
Period: Overall Study
Arm/Group | Specific Oral Tolerance Induction | Control
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Specific Oral Tolerance Induction | Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 10 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 7.033 (1.768) | 7.676 (3.203) | 7.354 (2.607)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  Italy | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Children That Achieved Total (40 ml) or Partial (Less Than 40 ml But at Least 10 ml) Tolerance to Raw Egg
Description: To evaluate the efficacy of a 6-month Specific Oral Tolerance Induction (SOTI) protocol in inducing tolerance (maximal dose of raw egg emulsion tolerated after 6 months) in children with severe IgE-mediated egg allergy and a history of at least 1 anaphylactic reaction after accidental exposure to egg.
Time Frame: baseline and 6 months
Measure: Number; unit: participants
Arm/Group | Specific Oral Tolerance Induction | Control
Number analyzed (Participants) | 10 | 10
participants | 9 | 0

2. Secondary Outcome: Changes in the Median Weal Diameter, Using Egg White SPTs, End-point SPT and PP
Description: Before and after SOTI, we evaluated the change in the median weal diameter in millimeters, using egg white SPTs, end-point SPT and PP.
Time Frame: Baseline and 6 months
Population: We were unable to calculate sample size because no quantitative data about the clinical outcome could be hypothesized. Indeed, the few reports of food causing allergy, the protocol, the way of SOTI administration and food doses administered yielded reported variable results. the analysis was per intention to treat
Measure: Median (Full Range); unit: mm diameter
Arm/Group | Specific Oral Tolerance Induction | Control
Number analyzed (Participants) | 10 | 10
mm diameter | 5 [4 to 13] | 10 [5.5 to 15]

ADVERSE EVENTS:
Time Frame: 6 month
Arm/Group | Specific Oral Tolerance Induction | Control
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Specific Oral Tolerance Induction (N=10) | Control (N=10)
Allergic reaction (Immune system disorders) | 10 (53) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No